CLINICAL TRIAL: NCT03831945
Title: An Exploratory Study of Combination Therapy With VRC-HIVMAB060-00-AB (VRC01) and 10-1074 in HIVInfected Individuals Undergoing Sequential Treatment Interruptions
Brief Title: Combination Therapy With VRC01 and 10-1074 in HIV-Infected Individuals Undergoing Sequential Treatment Interruptions
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: unable to recruit due to COVID pandemic
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 190048; 19-I-0048
Record Dates: First submitted 2019-02-05; First posted 2019-02-06 (Actual); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-08

CONDITIONS: HIV
Keywords: HIV Therapy; HIV Neutralizing Antibodies
MeSH Terms: interventions — VRC01 monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single infusion of VRC01 and 10-1074 (Active Comparator): Single infusion of 40 mg/kg VRC-HIVMAB060-00-AB (VRC01) in 100 mL of saline and 30 mg/kg of 10-1074 in 250 mL of saline when viral load is >/= 200 copies/mL in HIV-infected individuals undergoing antiretroviral treatment interruption.
  Interventions: Biological: VRC-HIVMAB060-00-AB (VRC01); Biological: 10-1074
- Single infusion of Normal Saline (Placebo Comparator): Single infusion of 100 mL and 250 mL of normal saline when viral load is >/= 200 copies/mL in HIV-infected individuals undergoing antiretroviral treatment interruption.
  Interventions: Biological: Normal Saline Placebo

INTERVENTIONS:
Biological: VRC-HIVMAB060-00-AB (VRC01) — VRC01 is a broadly neutralizing human mAb targeted against the HIV-1CD4 binding site. As single intravenous infusion of VRC01(40 mg/kg) plus10-1074 (30mg/kg) or placebo will be administered after the first analytical treatment interruption phase once the subject's plasma viremia is > or = 200 copies/mL.
  Arms: Single infusion of VRC01 and 10-1074
Biological: 10-1074 — 10-1074 is a recombinant, fully human mAb of the IgG1 lambda isotype that specifically binds to the base of the V3 loop within HIV-1 envelope gp-120. A single intravenous infusion of VRC01 (40 mg/kg) plus 10-1074 (30 mg/kg) or placebo will be administered after the first analytical treatment interruption phase once the subject's plasma viremia is > or = 200 copies/mL.
  Arms: Single infusion of VRC01 and 10-1074
Biological: Normal Saline Placebo — 2 sequential infusions of normal saline placebo in matching volumes to antibody infusions will be administered after the first analytical treatment interruption phase once the subject's plasma viremia is > or = 200 copies/mL.
  Arms: Single infusion of Normal Saline

SUMMARY:
Background:

A daily drug combination can keep human immunodeficiency virus (HIV) levels low for a long time. But if this combination antiretroviral therapy (ART) stops, HIV levels go back up. People can also develop resistance or permanent side effects. Researchers want to see if 2 new drugs can help control HIV when a person is not on ART.

Objective:

To see if VRC01 and 10-1074 are safe and control HIV when a person is not on ART.

Eligibility:

Adults 18-65 with HIV

Design:

All participants must agree to practice safer sex. Those who can get pregnant will have a pregnancy test every visit.

Participants will be screened with:

Physical exam

Medicine review

Blood and urine tests

Some participants may need to change their HIV medicine for a brief period of time during the study.

A few weeks later, participants will repeat screening tests and stop taking their HIV medicines.

Interruption phase 1: Participants will have blood tests every 2 weeks, and repeat screening tests every 4 weeks.

Treatment phase: Once their HIV reaches a certain level in the blood, participants will get the 2 study drugs or a salt water placebo. They will not know which they get. Each substance will be given through a thin tube in an arm vein for about 1 hour. Participants will restart their HIV medicines and repeat screening tests every 4 weeks.

Interruption phase 2: Once the level of HIV in the blood becomes undetectable for 3 months, participants will again stop taking their HIV medicines and have blood tests every 2 weeks to monitor the level of HIV in the blood.

Participants will restart their medicines by week 24. They will start sooner if they have certain symptoms or blood levels of HIV become too high. They will repeat most screening tests 3 times over 24 weeks.

DETAILED DESCRIPTION:
Recent advances in antibody cloning technologies have led to the development of a number of highly potent and human immunodeficiency virus (HIV)-specific broadly neutralizing monoclonal antibodies (bNAbs) from B cells of HIV-infected individuals. It has been shown that certain bNAbs can prevent acquisition of the virus, suppress viral replication, delay and/or prevent plasma viral rebound following treatment interruption in simian/human immunodeficiency virus (SHIV)-infected animals. Preliminary data from clinical trials indicates that bNAbs may delay plasma viral rebound following interruption of antiretroviral therapy (ART) and block cell-to-cell transmission of laboratory-adapted HIV in vitro.

In the above studies, suppression of plasma viremia was dependent on maintaining neutralizing serum levels of bNAbs via repeated intravenous (IV) infusions. A recent pre-clinical study in an acute SHIV-macaque model suggests a limited course of passive immunotherapy with two bNAbs (10-1074 and 3BNC117) given shortly after infection, can result in prolonged suppression of plasma viremia that is not dependent on the continuous presence of the bNAbs18. Based on CD8+ T cell depletion studies, it appears that the prolonged suppression of plasma viremia observed in these animals resulted from the induction of potent antiviral CD8+ T cell immunity by the short course bNAb treatment. The mechanism by which bNAb therapy could induce such a response is unclear but could involve the early formation of unique bNAb-SHIV immune complexes that subsequently induce an effective and durable T cell response to the virus.

In light of these encouraging preclinical outcomes, it is of considerable interest to investigate whether treatment with a single infusion of two bNAbs (VRC01 and 10-1074) which target different epitopes of HIV gp120 (CD4 binding site and V3 glycan, respectively), during transient plasma viremia can induce long-lasting anti-HIV immunity capable of controlling plasma viremia in the absence of ART.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. 18-65 years of age.
  2. HIV-1 infection and clinically stable.
  3. General good health and has an identified primary health care provider for medical management of HIV infection and is willing to maintain a relationship with a primary health care provider for medical management of HIV infection while participating in the study.
  4. CD4+ T cell count >450 cells/mm(3) at screening.
  5. Documentation of continuous ART treatment with suppression of plasma viral level below the lower limit of quantification (LLOQ) for the assay used for greater than or equal to 2 years. Individuals with blips (i.e., detectable viral levels on ART) prior to screening may be included provided they satisfy the following criteria:

     1. The blips are <400 copies/mL, and
     2. Succeeding viral levels return to levels below the limit of detection on subsequent testing.
  6. Laboratory values within pre-defined limits at screening:

     1. Absolute neutrophil count >1,000/mm(3).
     2. Hemoglobin levels >10.0 g/dL for men and >9.0 g/dL for women.
     3. Platelet count >100,000/mm(3).
     4. Estimated or a measured glomerular filtration rate >60 mL/min/1.73 m(2) as determined by the NIH Clinical Center (CC) laboratory.
     5. Aspartate aminotransferase (AST) and alanine transaminase (ALT) levels of <2.5 times upper limit of normal (ULN), direct bilirubin within the normal range for the NIH CC laboratory.
  7. Willingness to have samples stored for future research.
  8. Willingness to undergo analytical treatment interruption (ATI)
  9. Willingness for both male and female subjects to agree to use barrier protection methods or abstinence during the ATI phase of the study to decrease the risk of HIV transmission.

Reproductive Risks

Contraception: The effects of VRC01 and 10-1074 on the developing human fetus are unknown. For this reason, men and women of childbearing potential must agree to use adequate pregnancy prevention. This includes the use an effective method of contraception (i.e. condom with spermicide, diaphragm with spermicide, hormone-eluting intrauterine device (IUD), hormone-based contraceptive with condom) for the study duration. Subjects should also agree to use a male or female condom while off ART. Pregnancy prevention must be practiced continuously for the duration of study participation. Females of childbearing-age must have a negative pregnancy test result prior to receiving the infusions of VRC01 and 10-1074/placebo. During the course of the study, if a female subject, or the partner of a male subject suspects or in fact becomes pregnant, the affected subject should inform the study staff immediately, as well as the woman s primary care physician.

EXCLUSION CRITERIA:

1. Chronic hepatitis B, as evidenced by a positive test for hepatitis B surface antigen (HBsAg), or chronic hepatitis C virus (HCV) infection, as evidenced by a positive test for HCV RNA. Subjects with a positive test for HCV antibody and a negative test for HCV RNA are eligible.
2. HIV immunotherapy or HIV vaccine(s) received within 1 year prior to screening.
3. Any prior history of receiving 10-1074 or VRC01.
4. Any licensed or experimental non-HIV vaccination (e.g., hepatitis B, influenza, pneumococcal polysaccharide) received within 2 weeks prior to study enrollment.
5. Receipt of other investigational study agent within 28 days of enrollment.
6. Any active malignancy that may require systemic chemotherapy or radiation therapy.
7. Systemic immunosuppressive medications received within 3 months prior to enrollment (Exceptions: [1] corticosteroid nasal spray or inhaler; [2] topical corticosteroids for mild, uncomplicated dermatitis; or [3] oral/parenteral corticosteroids administered for non-chronic conditions not expected to recur [length of therapy less than or equal to 10 days, with completion in greater than or equal to 30 days prior to enrollment]).
8. History or other clinical evidence of:

   1. Significant or unstable cardiac or cerebrovascular disease (e.g., angina, congestive heart failure, recent stroke or myocardial infarction).
   2. Severe illness, malignancy, immunodeficiency other than HIV, or any other condition that, in the opinion of the investigator, would make the subject unsuitable for the study.
9. Active drug or alcohol use or any other pattern of behavior that, in the opinion of the investigator, would interfere with adherence to study requirements.
10. Pregnancy or breast-feeding at time of screening.
11. Documented multiclass antiretroviral drug resistance that, in the judgment of the investigator, would pose a risk of virologic failure should additional mutations develop during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Sneller, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Nishimura Y, Gautam R, Chun TW, Sadjadpour R, Foulds KE, Shingai M, Klein F, Gazumyan A, Golijanin J, Donaldson M, Donau OK, Plishka RJ, Buckler-White A, Seaman MS, Lifson JD, Koup RA, Fauci AS, Nussenzweig MC, Martin MA. Early antibody therapy can induce long-lasting immunity to SHIV. Nature. 2017 Mar 23;543(7646):559-563. doi: 10.1038/nature21435. Epub 2017 Mar 13. PMID 28289286
- [Background] Bar KJ, Sneller MC, Harrison LJ, Justement JS, Overton ET, Petrone ME, Salantes DB, Seamon CA, Scheinfeld B, Kwan RW, Learn GH, Proschan MA, Kreider EF, Blazkova J, Bardsley M, Refsland EW, Messer M, Clarridge KE, Tustin NB, Madden PJ, Oden K, O'Dell SJ, Jarocki B, Shiakolas AR, Tressler RL, Doria-Rose NA, Bailer RT, Ledgerwood JE, Capparelli EV, Lynch RM, Graham BS, Moir S, Koup RA, Mascola JR, Hoxie JA, Fauci AS, Tebas P, Chun TW. Effect of HIV Antibody VRC01 on Viral Rebound after Treatment Interruption. N Engl J Med. 2016 Nov 24;375(21):2037-2050. doi: 10.1056/NEJMoa1608243. Epub 2016 Nov 9. PMID 27959728
- [Background] Mendoza P, Gruell H, Nogueira L, Pai JA, Butler AL, Millard K, Lehmann C, Suarez I, Oliveira TY, Lorenzi JCC, Cohen YZ, Wyen C, Kummerle T, Karagounis T, Lu CL, Handl L, Unson-O'Brien C, Patel R, Ruping C, Schlotz M, Witmer-Pack M, Shimeliovich I, Kremer G, Thomas E, Seaton KE, Horowitz J, West AP Jr, Bjorkman PJ, Tomaras GD, Gulick RM, Pfeifer N, Fatkenheuer G, Seaman MS, Klein F, Caskey M, Nussenzweig MC. Combination therapy with anti-HIV-1 antibodies maintains viral suppression. Nature. 2018 Sep;561(7724):479-484. doi: 10.1038/s41586-018-0531-2. Epub 2018 Sep 26. PMID 30258136
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-I-0048.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 subjects were consented to protocol. 20 subjects started the study. Five subjects enrolled but not randomized due to the coronavirus disease 2019 (COVID 19) pandemic; one subject was lost to follow-up after enrollment, and one subjects not randomized due to hospitalization.
Period: Overall Study
Arm/Group | Single Infusion of VRC01 and 10-1074 | Single Infusion of Normal Saline
Started | 10 | 10
Completed | 3 | 4
Not Completed | 7 | 6
Not completed — Received study agent, never started second Analytical Treatment Interruption (ATI) due to COVID-19 | 4 | 4
Not completed — Received study agent, never started second analytical Treatment Interruption due to unprotected sex | 1 | 1
Not completed — Received study agent, second analytical treatment interruption (ATI) ended early due to COVID-19 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Infusion of VRC01 and 10-1074 | Single Infusion of Normal Saline | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 6 | 4 | 10
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Days From Start of the Second Treatment Interruption Until the Subject Meets Criteria to Restart ART
Description: Number of days from start of the second analytical treatment interruption (ATI) until the subject meets criteria to restart Antiretroviral Therapy (ART) before Week 16 [a confirmed >30% decline in baseline CD4+ T Cell count or an absolute CD4+ T Cell count in the setting of detectable HIV viremia (>40 copies/mL); a sustained (>4weeks) HIV RNA level of > 1000 copies/mL, or any HIV related symptoms or pregnancy.]
Time Frame: From start of second Analytical Treatment Interruption (ATI) until up to 16 weeks
Population: The analyses included all subjects who completed the second analytical treatment interruption phase. Because of safety concerns that stopping treatment for HIV during the current COVID-19 pandemic could increase the risk of getting severe COVID-19, the study was halted before sufficient participants had enrolled and completed the second analytical treatment interruption to accurately determine primary outcome
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Single Infusion of VRC01 and 10-1074 | Single Infusion of Normal Saline
Number analyzed (Participants) | 3 | 4
Days | 57 [50.5 to 59] | 63 [51.25 to 78.5]

2. Secondary Outcome: Percent of Participants With Grade 3 or Higher Related Adverse Events
Description: Percent of participants with grade 3 or higher adverse events, including serious adverse events, that were probably or definitely related to study agent
Time Frame: From the start of the initial infusion through follow-up phase week 24
Population: The analyses included all subjects who received at least one infusion of study agent
Measure: Number; unit: percentage of participants
Arm/Group | Single Infusion of VRC01 and 10-1074 | Single Infusion of Normal Saline
Number analyzed (Participants) | 10 | 10
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: After administration of study agent through follow-up phase week 24
Arm/Group | Single Infusion of VRC01 and 10-1074 | Single Infusion of Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Infusion of VRC01 and 10-1074 (N=10) | Single Infusion of Normal Saline (N=10)
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Infusion of VRC01 and 10-1074 (N=10) | Single Infusion of Normal Saline (N=10)
Proctitis (Gastrointestinal disorders) | 0 | 1
Salivary gland disorder (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Malaise (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Tenderness (General disorders) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gonorrhoea (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2
Skin infection (Infections and infestations) | 1 | 0
Syphilis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Echocardiogram abnormal (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Ageusia (Nervous system disorders) | 0 | 1
Anosmia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Depression (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Dental prosthesis user (Social circumstances) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT03831945/Prot_SAP_000.pdf